CLINICAL TRIAL: NCT02897687
Title: Project Rex Connect: The Utilization of an Online Social Network by an Interprofessional Team to Aid in Skill Acquisition for Patients With Autism Spectrum Disorders
Brief Title: Facebook for Social Skills Training in Autism: Project Rex Connect
Acronym: FBREX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00021530
Record Dates: First submitted 2016-08-12; First posted 2016-09-13 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Social Skills; Social Media
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Facebook Group (Experimental): Social skills training within an online group.
  Interventions: Behavioral: Facebook Group
- Book Club Group (Active Comparator): An in-person Book Club discussing material related to Autism Spectrum Disorder.
  Interventions: Behavioral: Book Club Group

INTERVENTIONS:
Behavioral: Facebook Group — A closed, invite-only group within Facebook facilitated by an interprofessional team that not only reinforces skills, but also aims to promote bonds and a sense of community and connectedness between participants.
  Arms: Facebook Group
Behavioral: Book Club Group — A topical book club group discussing Autism-related material conducted by a single healthcare professional.
  Arms: Book Club Group

SUMMARY:
Twelve participants were randomized to either a Facebook group or a book club group for six weeks. Data was collected on the participants social and behavioral function at both the start and the conclusion of the intervention.

DETAILED DESCRIPTION:
Research Design

The Project Rex team will randomize up to 12 subjects with Autism Spectrum Disorder who have completed the Project Rex Teen Treatment Group into either:

* (Group F) A closed, invite-only group within Facebook facilitated by an interprofessional team that not only reinforces skills, but also aims to promote bonds and a sense of community and connectedness between participants.

OR

* (Group B) A topical book club group conducted by a single healthcare professional.

Both treatment arms will be 8 weeks in duration. The interprofessional team for the Facebook arm of treatment will consist of one child and adolescent psychiatrist, one psychologist, two social workers and one medical student. The single professional conducting the book club activity will be a medical student. Parents will be required to help facilitate their child's participation in the study treatment. All study subjects will have completed the 8-week social skills introduction to social conversation Project Rex Teen group immediately prior to enrolling in either the Facebook arm (F) or the Book Club arm (B) of the study.

Upon completion of this treatment cycle, the study investigators will conduct an additional treatment cycle by randomizing two additional groups, each comprising up to 12 subjects with Autism Spectrum Disorder who have completed the 8-week Project Rex Teen Treatment Group into either Group F or Group B. The investigators will therefore enroll up to 24 total subjects in the study. The study is being divided into three cycles due to the limitation of recruiting only subjects who have completed the most recent round of the Project Rex teen program. Approval by the Medical University of South Carolina Institutional Review Board will be obtained before beginning this pilot study.

Study Procedure

Patients participating in the Project Rex Teen Group and their parents will be provided with written and verbal information about the opportunity to enroll in this study. This information will be disseminated to patients and parents after the completion of five of the total eight weeks of the Project Rex Teen Group. Patients and their parents will have opportunities to ask questions about the study with co-investigators after the sessions on week 6 and week 7. After the 8-week Project Rex teen group concludes, study co-investigators will be available to obtain informed consent from the parents of the subjects ages 12 to 17 years of age, and to obtain the assent of the respective subjects. The study investigators will also be available to obtain the informed consent of subjects who are age 18 to 20 years at the conclusion of the 8-week Project Rex Teen Group. The parents and subjects will have up to seven days after the conclusion of Week 8 of the Project Rex Teen Group to provide their informed consent and assent, respectively, for enrollment in the study.

Once parents and subjects have provided their informed consent/assent and the subjects are enrolled in the study, each subject will be randomized using REDCap into either Group F (Facebook arm) or Group B (Book Club Arm). Both subject groups and their parents will meet with for an information session about the study and their participation, which will be scheduled to occur within a week of the conclusion of Week 8 of the Project Rex Teen Program. Both treatment groups will meet on the same day and time, but will attend different information sessions located in different rooms within the Institute of Psychiatry.

All subjects who are assigned to the Facebook group and their parents will meet for a 90-minute group information session at Week 1, prior to the start of the Facebook treatment phase. These meetings will be conducted by the study investigators and will include a review of the study procedure, Facebook guidelines and Facebook terms and policy, privacy settings and data collection methods. The study investigators will directly support each subject in setting up their project Rex Facebook account and educating subjects about privacy settings. The study investigators will provide parents with education and training on the use of the Project Rex Facebook account and the maintenance of Project Rex Facebook account privacy settings to ensure that subjects are using the account appropriately and safely. At the conclusion of the Facebook information session, the subjects will be randomly assigned via lottery into two groups (1 & 2) for the purpose only of posting and responding to the discussion topic of the week.

All subjects and parents who are assigned to the Book Club group will meet for a 90-minute group information session at week 1, prior to the Book Club arm beginning. A study investigator will conduct this meeting and will provide a review of the study procedure, orient participants to the Book Club, review book club rules and expectations, and distribute the books.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Autism Spectrum Disorder
* Verbal

Exclusion Criteria:

* Non-verbal

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Improvements in social skills as assessed by Social Responsiveness Scale. | Week 1 and Week 8
Improvements in social skills as assessed by Social Skills Improvement System. | Week 1 and Week 8
Improvements in social skills as assessed by the Project Rex Parent Survey. | Week 1 and Week 8

SECONDARY OUTCOMES:
Participant satisfaction as assessed by the Project Rex Connect Participant Survey. | Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes